CLINICAL TRIAL: NCT04800341
Title: Collection of Medical Events Occurring During Long-term Follow-up in Patients Included in the European Sleep Apnea Data Base (ESADA)
Brief Title: Long-term Follow-up in Patients Included in the European Sleep Apnea Data Base (ESADA)
Acronym: ESADAfollow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.369; 2020-A03030-39 (Other: ID RCB)
Record Dates: First submitted 2020-12-07; First posted 2021-03-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Follow-up; Cardiovascular event; Metabolic event; Incident cancer; Death
MeSH Terms: conditions — Sleep Apnea Syndromes; Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients ESADA follow-up: Patients included in the ESADA European database and contacted by phone for the collection of cardiovascular and metabolic events, incident cancers and deaths, through a structured questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Structured questionnaire to collect cardiovascular and metabolic events, incident cancers and deaths that have occured, as weel as information on CPAP, through telephone interview.

SUMMARY:
The European database ESADA, containing data from more than 30,000 patients with very different severities of obstructive sleep apnea (OSA) syndrome, prospectively collects data from patients referred to academic sleep laboratories in many European countries (https://esada.med.gu.se/). Since 2007, Grenoble is one of the two French centers with Paris and is a very active participant in this European database for patient inclusion and data exploitation.

The first objective of the "ESADA Follow-up and outcomes" project is to collect cardiovascular events during the follow-up of patients in the European database through telephone interviews and a structured questionnaire. Other objectives are to collect metabolic events, incident cancers and deaths in the same population using the same mean.

An additional objective is to assess the impact of continuous positive airway pressure (CPAP, the reference treatment for OSA) on the occurrence of cardiovascular and metabolic events and incident cancers, as this is still discussed in the literature.

DETAILED DESCRIPTION:
The European database ESADA prospectively collects data from patients referred to academic sleep laboratories in many European countries (https://esada.med.gu.se/). Since 2007, Grenoble is one of the two French centers with Paris and is a very active participant in this European database for patient inclusion and data exploitation. A partnership agreement exists between University Hospital Grenoble (CHUGA) and ESADA for the reuse of CHUGA data. The data collected at CHUGA as part of the ESADA-Follow-up and outcomes questionnaire are also collected in the other European centers and will be centralized at the level of the coordinating center.

ESADA currently contains data from more than 30,000 patients with very different severities of obstructive sleep apnea (OSA) syndrome. One of the main limitations of this cohort is the relatively limited amount of information concerning the long-term follow-up of the patients included in the registry.

The first objective of the "ESADA Follow-up and outcomes" project is to collect cardiovascular events during the follow-up of patients in the European database through telephone interviews and a structured questionnaire. Other objectives are to collect metabolic events, incident cancers and deaths in the same population using the same mean.

An additional objective at the end of this data collection is to aggregate the follow-up data of more than 10,000 patients from all participating European centers to assess the impact of continuous positive airway pressure (CPAP, the reference treatment for OSA) on the occurrence of cardiovascular and metabolic events and incident cancers, as this is still discussed in the literature.

ELIGIBILITY:
Inclusion Criteria:

* already included in the ESADA European database

Exclusion Criteria:

* refusal to participate

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sleep apnea patients included in the ESADA European database
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiovascular events | up to 15 years
  Prevalence of cardiovascular events during the follow-up of patients included in the ESADA European database, through a structured questionnaire.
Prevalence of metabolic events | up to 15 years
  Prevalence of metabolic events during the follow-up of patients included in the ESADA European database, through a structured questionnaire.
Prevalence of incident cancers | up to 15 years
  Prevalence of incident cancers during the follow-up of patients included in the ESADA European database, through a structured questionnaire.
Prevalence of deaths | up to 15 years
  Prevalence of deaths during the follow-up of patients included in the ESADA European database, through a structured questionnaire.

SECONDARY OUTCOMES:
Effect of CPAP treatment on the cardiovascular events occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the ESADA European database to determine its impact on the cardiovascular events occurrence.
Effect of CPAP treatment on the metabolic events occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the ESADA European database to determine its impact on the metabolic events occurrence.
Effect of CPAP treatment on the incident cancers occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the ESADA European database to determine its impact on the incident cancers occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No